CLINICAL TRIAL: NCT02810444
Title: An Open-label, Prospective, Multicenter Study Investigating Clinical Efficacy, Safety, and Pharmacokinetic Properties of the Human Normal Immunoglobulin for Intravenous Administration BT595 as Replacement Therapy in Patients With Primary Immunodeficiency Disease (PID)
Brief Title: Study to Investigate Efficacy, Safety and Pharmacokinetics of BT595 in Subjects With PID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotest (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 991; 2015-003652-52 (EudraCT Number)
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Primary Immunodeficiency Disease
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BT595 (Experimental): Subjects received BT595 (100 mg/mL human normal immunoglobulin) at doses between 0.2 and 0.8 g per kg body weight (bw) (2 to 8 mL/kg bw), either at a Q3W or Q4W schedule, The initial doses and dosage interval had to be consistent with the subject's prestudy IVIg treatment.
  Interventions: Biological: IgG Next Generation (BT595)

INTERVENTIONS:
Biological: IgG Next Generation (BT595)
  Other Names: Immune Globulin Intravenous (Human), 10% Liquid

SUMMARY:
This Phase III clinical study is to test efficacy, safety and pharmacokinetics of BT595 in treating patients with Primary Immunodeficiency (PID)

ELIGIBILITY:
Criteria for inclusion:

1. Written informed consent/assent obtained from subjects/subjects' parent(s) or legally acceptable representative indicating that they understood the purpose of, and procedures required for the study and are willing to participate in it.
2. Male or female, aged 2 through 75 years, inclusive.
3. Diagnosis of PID with impaired antibody production, ie:

   - Diagnosis of common variable immunodeficiency (CVID) as defined by the European Society for Immunodeficiencies (ESID)/Pan American Group for Immunodeficiency (PAGID) diagnostic criteria.

   Or

   - X-linked agammaglobulinaemia (XLA) as defined by ESID/PAGID diagnostic criteria.
4. Established replacement therapy with any immunoglobulin for intravenous administration (IVIg) reference preparation during the previous 6 months, including documentation of IgG trough levels.
5. Established replacement therapy with a single IVIg reference preparation for ≥3 months prior to treatment start with BT595 at a 3 week (Q3W) or 4 week (Q4W) schedule with a constant IVIg dose that did not change by ±20% of the mean dose, regular dosage intervals, and at least 1 IgG trough level of ≥5 g/L during the previous 3 months.

Criteria for exclusion:

1. Pregnancy or unreliable contraceptive measures or lactation period (females only).
2. Known intolerance to immunoglobulins or comparable substances (eg, vaccination reaction).
3. Known intolerance to proteins of human origin or known allergic reactions to components of the study product.
4. Participation in another clinical study within 30 days before entering the study or during the study and/or previous participation in this study.
5. Employee or direct relative of an employee of the contract research organization, the study site, or Biotest.
6. Acquired medical conditions known to cause secondary immune deficiency, such as chronic lymphatic leukemia, lymphoma, multiple myeloma, as well as protein losing enteropathies and hypoalbuminemia.
7. Other medical condition, laboratory finding, or physical examination finding that precludes participation.
8. Recent febrile illness that precludes or delays participation.
9. Active infection and receiving antibiotic therapy for the treatment of this infection at the time of screening. Note: if the subject was deemed to be a screen failure due to a nonserious active infection requiring antibiotic therapy, the subject may have been rescreened after the initial screening.
10. Therapy with systemic steroids or other immunosuppressant drugs at the time of enrollment (current daily use of corticosteroids, ie, >10 mg prednisone equivalent/day for >30 days. Intermittent corticosteroid use during the study was allowable, if medically necessary).
11. History of thrombotic events (including myocardial infarction, cerebral vascular accident [including stroke], pulmonary embolism, and deep vein thrombosis) within the 6 months before treatment start with BT595 or the presence of significant risk factors for thrombotic events.
12. Therapy with live-attenuated virus vaccines within 3 months before start of the study.
13. Selective, absolute immunoglobulin A (IgA) deficiency or known antibodies to IgA.
14. Positive diagnosis of hepatitis B or hepatitis C.
15. Positive human immunodeficiency virus (HIV) test.
16. History of drug or alcohol abuse within the 12 months before treatment start with BT595.
17. Inability or lacking motivation to participate in the study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gergely Krivan, MD, Principal Investigator — Egyesitett Szent Istvan es Szent Laszlo Korhaz, Budapest, Hungary
Locations (19):
- United States (9):
  - Investigational site # 0104, Birmingham, Alabama
  - Investigational site # 0116, Los Angeles, California
  - Investigational site # 0103, Centennial, Colorado
  - Investigational site # 0114, Thornton, Colorado
  - Investigational site # 0111, Chicago, Illinois
  - Investigational site # 0106, South Bend, Indiana
  - Investigational site # 0105, Toledo, Ohio
  - Investigational site #0115, Memphis, Tennessee
  - Investigational Site # 0102, Dallas, Texas
- Germany (3):
  - Investigational site # 4902, Frankfurt am Main
  - Investigational site # 4904, Freiburg im Breisgau
  - Investigational site #4905, Leipzig
- Hungary (3):
  - Investigational site # 3602, Budapest
  - Investigational Site # 3605, Miskolc
  - Investigational site #3603, Nyíregyháza
- Russia (2):
  - Investigational site # 0702, Moscow
  - Investigational site # 0704, Yekaterinburg
- Spain (2):
  - Investigational site # 3403, Barcelona
  - Investigational site # 3405, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krivan G, Borte M, Harris JB, Lumry WR, Aigner S, Lentze S, Staiger C. Efficacy, safety and pharmacokinetics of a new 10% normal human immunoglobulin for intravenous infusion, BT595, in children and adults with primary immunodeficiency disease. Vox Sang. 2022 Oct;117(10):1153-1162. doi: 10.1111/vox.13337. Epub 2022 Aug 9. PMID 35944615
- [Result] Krivan G, Borte M, Soler-Palacin P, Church JA, Csurke I, Harris JB, Lieberman JA, Melamed IR, Moy JN, Simon R, Aigner S, Lentze S, Staiger C. BT595, a 10% Human Normal Immunoglobulin, for Replacement Therapy of Primary Immunodeficiency Disease: Results of a Subcohort Analysis in Children. J Clin Immunol. 2023 Apr;43(3):557-567. doi: 10.1007/s10875-022-01397-0. Epub 2022 Nov 16. PMID 36383294

RESULTS

PARTICIPANT FLOW:
Groups:
- BT595: Subjects received BT595 (100 mg/mL human normal immunoglobulin) at doses between 0.2 and 0.8 g per kg body weight (bw) (2 to 8 mL/kg bw), either at a Q3W or Q4W schedule. The initial doses and dosage interval had to be consistent with the subject's prestudy IVIg treatment.
Period: Overall Study
Arm/Group | BT595
Started | 81 (as defined by protocol)
Treatment Started | 67
Completed | 60
Not Completed | 21
Not completed — Screen Failures | 14
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | BT595
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 44
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 28
  United States | 21
  Germany | 4
  Spain | 3
  Russia | 11

OUTCOME MEASURES:

1. Primary Outcome: Rate of Acute Serious Bacterial Infections
Description: The primary efficacy endpoint was the rate of acute serious bacterial infections, ie, the mean number of acute serious bacterial infections [SBIs as defined by EMA and FDA] per subject-year.
Time Frame: approx. 12 month treatment period
Population: The primary analysis intended to demonstrate that the SBI rate (upper limit of the 1-sided 99% CI) was <1.0 per subject-year in the overall FAS
Measure: Number; unit: SBI rate per subject-year
Arm/Group | BT595
Number analyzed (Participants) | 67
SBI rate per subject-year | 0.015

2. Secondary Outcome: IgG Trough Levels (Total IgG) Before Each Infusion
Description: Total IgG levels [g/L] before each infusion, mean (SD)
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | BT595
Number analyzed (Participants) | 67
g/L
  Screening, Q4W: number analyzed (Participants) | 55
  Screening, Q4W | 8.467 (3.4562)
  Baseline, Q4W: number analyzed (Participants) | 55
  Baseline, Q4W | 7.824 (2.7705)
  Infusion 1 (Week 0), Q4W: number analyzed (Participants) | 55
  Infusion 1 (Week 0), Q4W | 7.824 (2.7705)
  Infusion 2 (Week 4), Q4W: number analyzed (Participants) | 50
  Infusion 2 (Week 4), Q4W | 8.278 (2.5919)
  Infusion 3 (Week 8), Q4W: number analyzed (Participants) | 51
  Infusion 3 (Week 8), Q4W | 8.246 (2.3970)
  Infusion 4 (Week 12), Q4W: number analyzed (Participants) | 51
  Infusion 4 (Week 12), Q4W | 8.410 (2.2998)
  Infusion 5 (Week 16), Q4W: number analyzed (Participants) | 52
  Infusion 5 (Week 16), Q4W | 8.634 (3.4997)
  Infusion 6 (Week 20), Q4W: number analyzed (Participants) | 51
  Infusion 6 (Week 20), Q4W | 8.203 (2.2912)
  Infusion 7 (Week 24), Q4W: number analyzed (Participants) | 52
  Infusion 7 (Week 24), Q4W | 8.298 (2.3822)
  Infusion 8 (Week 28), Q4W: number analyzed (Participants) | 50
  Infusion 8 (Week 28), Q4W | 8.308 (2.1087)
  Infusion 9 (Week 32), Q4W: number analyzed (Participants) | 52
  Infusion 9 (Week 32), Q4W | 8.410 (2.2353)
  Infusion 10 (Week 36), Q4W: number analyzed (Participants) | 52
  Infusion 10 (Week 36), Q4W | 8.264 (2.2994)
  Infusion 11 (Week 40), Q4W: number analyzed (Participants) | 51
  Infusion 11 (Week 40), Q4W | 8.181 (2.1706)
  Infusion 12 (Week 44), Q4W: number analyzed (Participants) | 52
  Infusion 12 (Week 44), Q4W | 8.336 (2.0893)
  Infusion 13 (Week 48), Q4W: number analyzed (Participants) | 49
  Infusion 13 (Week 48), Q4W | 8.479 (2.3571)
  Infusion 14 (Week 52), Q4W: number analyzed (Participants) | 48
  Infusion 14 (Week 52), Q4W | 8.437 (2.1703)
  Infusion 15 (extra dose administered), Q4W: number analyzed (Participants) | 4
  Infusion 15 (extra dose administered), Q4W | 8.950 (0.6608)
  Follow-up, Q4W: number analyzed (Participants) | 49
  Follow-up, Q4W | 8.461 (2.2248)
  Screening, Q3W: number analyzed (Participants) | 12
  Screening, Q3W | 10.238 (2.4700)
  Baseline, Q3W: number analyzed (Participants) | 12
  Baseline, Q3W | 10.064 (2.6829)
  Infusion 1 (Week 0), Q3W: number analyzed (Participants) | 11
  Infusion 1 (Week 0), Q3W | 10.261 (2.7216)
  Infusion 2 (Week 3), Q3W: number analyzed (Participants) | 11
  Infusion 2 (Week 3), Q3W | 10.422 (2.9521)
  Infusion 3 (Week 6), Q3W: number analyzed (Participants) | 11
  Infusion 3 (Week 6), Q3W | 10.509 (2.9857)
  Infusion 4 (Week 9), Q3W: number analyzed (Participants) | 11
  Infusion 4 (Week 9), Q3W | 10.050 (3.0155)
  Infusion 5 (Week 12), Q3W: number analyzed (Participants) | 11
  Infusion 5 (Week 12), Q3W | 10.267 (3.2398)
  Infusion 6 (Week 15), Q3W: number analyzed (Participants) | 11
  Infusion 6 (Week 15), Q3W | 10.026 (3.2135)
  Infusion 7 (Week 18), Q3W: number analyzed (Participants) | 9
  Infusion 7 (Week 18), Q3W | 10.032 (2.2755)
  Infusion 8 (Week 21), Q3W: number analyzed (Participants) | 10
  Infusion 8 (Week 21), Q3W | 10.268 (2.7719)
  Infusion 9 (Week 24), Q3W: number analyzed (Participants) | 10
  Infusion 9 (Week 24), Q3W | 9.889 (2.1752)
  Infusion 10 (Week 27), Q3W: number analyzed (Participants) | 10
  Infusion 10 (Week 27), Q3W | 10.343 (2.2324)
  Infusion 11 (Week 30), Q3W: number analyzed (Participants) | 10
  Infusion 11 (Week 30), Q3W | 10.188 (2.6981)
  Infusion 12 (Week 33), Q3W: number analyzed (Participants) | 10
  Infusion 12 (Week 33), Q3W | 10.427 (2.7320)
  Infusion 13 (Week 36), Q3W: number analyzed (Participants) | 9
  Infusion 13 (Week 36), Q3W | 10.087 (2.6267)
  Infusion 14 (Week 39), Q3W: number analyzed (Participants) | 10
  Infusion 14 (Week 39), Q3W | 10.245 (2.4434)
  Infusion 15 (Week 42), Q3W: number analyzed (Participants) | 10
  Infusion 15 (Week 42), Q3W | 10.539 (2.2490)
  Infusion 16 (Week 45), Q3W: number analyzed (Participants) | 10
  Infusion 16 (Week 45), Q3W | 10.045 (2.7147)
  Infusion 17 (Week 48), Q3W: number analyzed (Participants) | 10
  Infusion 17 (Week 48), Q3W | 9.877 (2.0190)
  Infusion 18 (Week 51), Q3W: number analyzed (Participants) | 9
  Infusion 18 (Week 51), Q3W | 10.412 (2.4921)
  Follow-up, Q3W: number analyzed (Participants) | 10
  Follow-up, Q3W | 10.415 (2.6176)

3. Secondary Outcome: Rate of Any Infections
Description: The annual rate of infections was calculated as the number of all infections (serious plus nonserious) per subject-year
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Number; unit: infections per subject-year
Arm/Group | BT595
Number analyzed (Participants) | 67
infections per subject-year | 2.80

4. Secondary Outcome: Rate of Nonserious Infections
Description: The annual rate of nonserious infections was calculated as the number of nonserious infections per subject-year
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Number; unit: infections per subject-year
Arm/Group | BT595
Number analyzed (Participants) | 67
infections per subject-year | 2.74

5. Secondary Outcome: Time to Resolution of Infections
Description: Time to resolution of infections (days) was calculated as infection stop date - infection start date +1.
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Median (Full Range); unit: days
Arm/Group | BT595
Number analyzed (Participants) | 67
days | 7.0 [7.0 to 8.0]

6. Secondary Outcome: Antibiotic Treatment Information
Description: Median (min-max) number of days on antibiotics treatment per subject
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Median (Full Range); unit: days
Arm/Group | BT595
Number analyzed (Participants) | 67
days | 6.0 [0 to 409]

7. Secondary Outcome: Rate of Time Lost From School/Work Due to Infections
Description: Annual rates of the number of days subjects are not able to attend school/work due to infections and their treatment will be calculated per subject-year.
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Number; unit: days per subject-year
Arm/Group | BT595
Number analyzed (Participants) | 67
days per subject-year | 4.32

8. Secondary Outcome: Hospitalization / Hospitalization Due to Infection
Description: Annual rates of the number of days of hospitalization (any hospitalization/ hospitalization due to infection) will be calculated per subject-year.
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Number; unit: days per subject-year
Arm/Group | BT595
Number analyzed (Participants) | 67
days per subject-year
  Any Hospitalization | 0.70
  Hospitalization due to Infection | 0.36

9. Secondary Outcome: Fever Episodes
Description: The number of days with episodes of fever will be calculated as the number of fever episodes per subject-year. Fever is defined as a body temperature ≥38°C (≥100.4°F).
Time Frame: approx. 12 month treatment period
Population: Full analysis set
Measure: Number; unit: days per subject-year
Arm/Group | BT595
Number analyzed (Participants) | 67
days per subject-year | 1.69

ADVERSE EVENTS:
Time Frame: During treatment phase until Follow-up visit approx. 1 year
Arm/Group | BT595
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 9/67
Other Adverse Events (participants affected / at risk) | 63/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT595 (N=67)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — related TEAE
Hepatitis toxic (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) — related TEAE
Anal abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT595 (N=67)
Diarrhoea (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 6 (10)
Bronchitis (Infections and infestations) | 8 (12)
Conjunctivitis (Infections and infestations) | 4 (6)
Influenza (Infections and infestations) | 6 (6)
Nasopharyngitis (Infections and infestations) | 16 (24)
Pharyngitis (Infections and infestations) | 7 (8)
Sinusitis (Infections and infestations) | 8 (11)
Upper respiratory tract infection (Infections and infestations) | 13 (24)
Urinary tract infection (Infections and infestations) | 6 (8)
Viral upper respiratory tract infection (Infections and infestations) | 7 (7)
Extra dose administered (Injury, poisoning and procedural complications) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Headache (Nervous system disorders) | 17 (41)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT02810444/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT02810444/SAP_001.pdf